CLINICAL TRIAL: NCT04223739
Title: Comparison of Two Strategies for the Management of Atrial Fibrillation After Cardiac Surgery : a Randomized Multicenter Clinical Trial
Brief Title: Comparison of Two Strategies for the Management of Atrial Fibrillation After Cardiac Surgery
Acronym: FAAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A00763-54
Record Dates: First submitted 2019-12-13; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: Cardiac Surgery; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — landiolol; Amiodarone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol (Active Comparator): Landiolol infusion starting at 2.5 µg/kg/min and titrating up to 80µg/kg/min with a heart rate goal of under 90 bpm.
  Interventions: Drug: Landiolol
- Amiodarone (Active Comparator): Amiodarone bolus of 5-7 mg/kg in 1 hour, followed by an infusion of 1g/day until conversion to sinus rhythm.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Landiolol — Landiolol infusion with incremental doses (range from 2,5µg/kg/min to 80 µg/kg/min) with go of heart rate < 90 bpm. Doses are modified every 10 minutes if necessary.
  Once heart rate goal is obtained, switch to an oral dose of Bisoprolol.
  Other Names: Rapibloc
  Arms: Landiolol
Drug: Amiodarone — Amiodarone loading dose of 5-7 mg/kg in 1 hour followed by an infusion of 1 g/day until conversion to sinus rhythm. Once sinus rhythm is obtained, switch to an oral dose of 200mg/day
  Other Names: Cordarone
  Arms: Amiodarone

SUMMARY:
Postoperative atrial fibrillation is a common complication after cardiac surgery with a rate of 30%. However, management of postoperative atrial fibrillation is controversial. Two strategies are recommended : heart rate control using a betablocker or rhythm control with amiodarone.

Landiolol is a new-generation beta-blocker with a short half-life, which was approved by the Haute Autorité de Santé to be used in perioperative supra-ventricular tachycardias.

Only one study compared landiolol to amiodarone in the perioperative setting, with a better hemodynamic tolerance and a higher rate of conversion to sinus rhythm with landiolol. However this was a single-center and retrospective study.

The aim of our multicenter randomized study is to compare the effectiveness of landiolol in reducing atrial fibrillation to sinus rhythm compared to amiodarone in the postoperative period after cardiac surgery.

DETAILED DESCRIPTION:
Randomized clinical study comparing landiolol and amiodarone for treatment of atrial fibrillation following cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in the cardiac ICU after having undergone cardiac surgery (CABG, aortic valve or ascending aortic root replacement or a combination of both)
* New onset of atrial fibrillation lasting more than 30 minutes in the postoperative period after cardiac surgery
* French speaking patients
* Written consent
* Patients with social security insurance

Exclusion Criteria:

* Hemodynamic instability requiring electrical cardioversion of atrial fibrillation
* Sepsis
* Bradyarrythmia (< 90/min)
* Patients requiring inotropes in the postoperative period
* Patient with pre-existing atrial fibrillation
* Patient with anticoagulant therapy before surgery
* Contraindication to amiodarone or beta-blockers
* Urgent surgery (< 24h), ventricular assist device, heart transplant, TAVR, mechanical valve, mitral or tricuspid valve replacement.
* No written consent
* Pregnant women,
* Underaged patients (<18 years old)
* Patients not able to give consent (curators, patients deprived of public rights)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in sinus rhythm 48 hours after the onset of atrial fibrillation immediate postoperative period after cardiac surgery | Day 2 after onset of atrial fibrillation
  Percentage of patients in sinus rhythm 48 hours after the onset of atrial fibrillation immediate postoperative period after cardiac surgery

SECONDARY OUTCOMES:
Haemodynamic side effects (hypotension, bradycardia) | Day 8 after onset of atrial fibrillation and through hospital discharge, an average of 14 days
  Haemodynamic side effects (hypotension, bradycardia)
Length of hospital stay | Day 8 after onset of atrial fibrillation and through hospital discharge, an average of 14 days
  Length of stay in the hospital from randomisation to hospital discharge
Rate of thrombo-embolic events | 2 months postsugery and 1 year postsurgery
  Rate of stroke or ischemic embolism
Quality of life evaluated by the EQ 5D 3L questionnaire | 2 months postsurgery and 1 year postsurgery
  Quality of life as evaluated by the EQ 5D 3L questionnaire
Rate of atrial fibrillation recurrence | 2 months postsurgery and 1 year postsurgery
  Percentage of patients having a recurrence of atrial fibrillation after the initial conversion to sinus rythm in the postoperative period
Severe hemorrhagic complications due to anticoagulant therapy, as defined by the Haute Autorité de Santé | 2 months postsurgery and 1 year postsurgery
  Hemorrhagic complications requiring surgery or interventional radiology Hemorrhagic complications responsible of hemodynamic instability (Systolic Arterial Pressure < 90 mmHg, or drop of more than 40 mmHg or Mean Arterial Pressure < 65 mmHg or signs of shock) Life threatening hemorrhagic complications (intracerebral, intramedullar or intraocular hemorrhage, hemothorax, abdominal hemorrhage, deep muscular hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Caspersen, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, Calvados, France

REFERENCES:
- [Derived] Caspersen E, Guinot PG, Rozec B, Oilleau JF, Fellahi JL, Gaudard P, Lorne E, Mahjoub Y, Besnier E, Moussa MD, Mongardon N, Hanouz JL, Briant AR, Paul LPS, Tomadesso C, Parienti JJ, Descamps R, Denisenko A, Fischer MO; ARCOTHOVA Group. Comparison of landiolol and amiodarone for the treatment of new-onset atrial fibrillation after cardiac surgery (FAAC) trial: study protocol for a randomized controlled trial. Trials. 2023 May 25;24(1):353. doi: 10.1186/s13063-023-07353-6. PMID 37226174